CLINICAL TRIAL: NCT06504550
Title: Comparison Between Schroth AND Klapp Method On Postural Stability AND Trunk Rotation Angle In CP Children With Scoliosis
Brief Title: Comparison Between Schroth and Klapp Method in CP Children With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0779
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy; Scoliosis
Keywords: Cerebral Palsy; Klapp; Postural Stability; Schroth; Scoliosis; Trunk Rotation Angle
MeSH Terms: conditions — Cerebral Palsy; Scoliosis

STUDY DESIGN:
Intervention Model Description: It will be Randomized clinical trial in which non probability convinient sampling will be used.Two groups of 8 to 12 years of age will be formed in which participants will be randomly divided.In Group A Schroth exercises will be conducted that consist of passive and active postural auto-correction exercises done repeatedly and based on kinesthetic and sensorimotor principles.In Group B Klapp group will be treated with klapp exercises. In each session, a sequence of 8 postures of Klapp method will be carried out
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth Exercise. Group A receive Schroth Exercises. (Experimental): Group A: Schroth Group (SG). The patients in the Schroth exercise group will start their exercise program under physiotherapist supervision. Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks. These exercises include spinal elongation, de-rotation, de-flexion, stretching, strengthening to maintain vertebral alignment.The participants will be asked to combine these exercises with their daily living activities (ADLs).During the Schroth exercises, rice bags, foam blocks, a stool, and long sticks will be used to adjust the posture and give passive support.Exercises are progressed from lying, sitting, or standing positions and from most to least passive support per a review of the quality of the performance.Decreasing the amount or degree of passive support, changing the patient's position, and adjusting the sets and repetitions of exercises will depend on the patient's improvement in exercise performance
  Interventions: Other: Schroth Exercises
- Klapp Exercise. Group B receive Klapp Exercises. (Experimental): Group B: Klapp group (KG). The patients in the Klapp exercise group will be treated with supervised klapp exercises.Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks.In each session, a sequence of 8 postures of Klapp Exercises will be carried out.Each posture will be maintained for 4-5 minutes with rest breaks when needed.Positions that will be held are: 1) Lateral crawl, 2) Horizontal sliding, 3) Crawl posture near the ground, 4) Bunny hopping, 5) Arm turn, 6) Big arch, 7) Lateral crawl near the ground, 8) Big curve
  Interventions: Other: Klapp Exercises

INTERVENTIONS:
Other: Schroth Exercises — The patients in the Schroth exercise group will start their exercise program under physiotherapist supervision.Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks.These exercises include spinal elongation, de-rotation, de-flexion, stretching, strengthening exercises to maintain vertebral alignment.The participants will be asked to combine these exercises with their daily living activities (ADLs).During the Schroth exercises, rice bags, foam blocks, a stool, and long sticks will be used to adjust the posture and give passive support.Exercises are progressed from lying, sitting, or standing positions and from most to least passive support per a review of the quality of the performance.Decreasing the amount or degree of passive support, changing the patient's position, and adjusting the sets and repetitions of exercises will depend on the patient's improvement in exercise performance
  Arms: Schroth Exercise. Group A receive Schroth Exercises.
Other: Klapp Exercises — The patients in the Klapp exercise group will be treated with supervised klapp exercises. Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks.In each session, a sequence of 8 postures of Klapp Exercises will be carried out. Each posture will be maintained for 4-5 minutes with rest breaks when needed.Positions that will be held are: 1) Lateral crawl, 2) Horizontal sliding, 3) Crawl posture near the ground, 4) Bunny hopping, 5) Arm turn, 6) Big arch, 7) Lateral crawl near the ground, 8) Big curve
  Arms: Klapp Exercise. Group B receive Klapp Exercises.

SUMMARY:
Cerebral palsy, which occurs in two to three out of 1,000 live births, has multiple etiologies resulting in brain injury that affects movement, posture, and balance. Approximately one-third of children with CP are non-ambulant and subsequently spend prolonged periods of time in sitting or lying. Non-ambulatory patients with cerebral palsy (CP) bear a high risk of developing simultaneous progressive scoliotic spine deformities, loss of sitting balance and hip subluxation/dislocation.Treatments for the Spinal deformities associated with cerebral palsy are Schroth method. It is a scoliosis-specific exercise approach that uses postural, scoliosis-specific sensorimotor exercises. While another treatment approach Klapp method aimed to stretch and strengthen muscles by all fours positions, easily applied and that can be used in small groups.

A Randomized clinical trial will be conducted through convenient sampling. Inclusion criteria of this study is age between 8 to 12 years of either gender, with GMFCS level I and II and Trunk rotation angle (ATR) > 4 degree, who are able to understand and follow verbal instructions. Those patients who has been prescribed brace treatment, has scheduled or undergone any corrective surgical treatment of the spine before or during data collection process will be excluded. Patients who are unable to participate, or are reluctant to receive treatment are excluded. Study will be conducted on 22 patients who will be randomly allocated into two groups. One group will receive Schroth exercises. It consists of passive and active postural auto-correction exercises done repeatedly and based on kinesthetic and sensorimotor principles. While the other group with Klapp method includes stretching and strengthening muscles by all fours positions. Bunnell's scoliometer, Adams forward bend test, and Posture and postural ability scale (PPAS) will be used as outcome measure.

DETAILED DESCRIPTION:
Group A is Schroth Group (SG). The patients in the Schroth exercise group will start their exercise program under physiotherapist supervision. Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks. Schroth exercises will be performed in an asymmetric position to maximize correction to achieve trunk symmetry. These exercises include spinal elongation, de-rotation, de-flexion, stretching, strengthening and rotational breathing exercises to maintain vertebral alignment. The participants will be asked to combine these exercises with their daily living activities (ADLs). During the Schroth exercises, rice bags, foam blocks, a stool, and long sticks will be used to adjust the posture and give passive support. Exercises are progressed from lying, sitting, or standing positions and from most to least passive support per a review of the quality of the performance. Decreasing the amount or degree of passive support, changing the patient's position, and adjusting the sets and repetitions of exercises will depend on the patient's improvement in exercise performance Group B is Klapp group (KG).The patients in the Klapp exercise group will be treated with supervised klapp exercises. Exercise treatment program will consist of 18 sessions, 30 minutes each session, three times a week, for 6 weeks. In each session, a sequence of 8 postures of Klapp Exercises will be carried out. Each posture will be maintained for 4-5 minutes with rest breaks when needed. Positions that will be held are: 1) Lateral crawl, 2) Horizontal sliding, 3) Crawl posture near the ground, 4) Bunny hopping, 5) Arm turn, 6) Big arch, 7) Lateral crawl near the ground, 8) Big curve

ELIGIBILITY:
Inclusion Criteria:

* 8 to 12 years of age
* Either gender.
* The level of gross motor function between levels I and II in accordance with the gross motor function classification system (GMFCS) .
* Angle of Trunk Rotation (ATR) > 4 degree .
* Ability to understand and follow verbal instructions

Exclusion Criteria:

* Patients will be excluded if they have had been prescribed brace treatment
* Has received any previous corrective or surgical treatment of the spine
* Unable to participate, or are reluctant to receive treatment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Posture and Postural Ability Scale (PPAS) | 6 weeks
  An assessment tool for measuring the quality of postures as well as classifying the ability to maintain and manipulate postures.The Posture and Postural Ability Scale (PPAS) is used to assess supine, prone, lying and sitting posture in the frontal and sagittal planes. The scale ranges from full symmetry to total asymmetry. Similarly, their ability to change or maintain position was rated according to the levels of PPAS ranging from "Able to move into and out of position independently" (level 7) to "Unplaceable in an aligned position" (level 1).The PPAS has excellent inter-rater reliability and validity for children and adults with CP
Bunnell's Scoliometer | 6 weeks
  Trunk rotation angle (ATR) will be evaluated using Bunnell's scoliometer and Adam's forward bend test. For patients with scoliosis, a landmark for measuring the angle of trunk rotation will be marked on the protruding area during the forward bending test using a scoliometer. For measuring the angle of trunk rotation of scoliosis patient, in order to set the reference point of the scoliometer, the scoliometer is placed on the floor and focused. In the forward bending test, the angle of trunk rotation is measured using a scoliometer on the area to be measured marked with a sticker. The measured value will be read and recorded. The inter-rater reliability according to the measurement method with Scoliometer measurement method 0.971. The scoliometer measurement method has the highest validity (r=0.976)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Khaliq, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agustsson A, Sveinsson T, Pope P, Rodby-Bousquet E. Preferred posture in lying and its association with scoliosis and windswept hips in adults with cerebral palsy. Disabil Rehabil. 2019 Dec;41(26):3198-3202. doi: 10.1080/09638288.2018.1492032. Epub 2018 Jul 16. PMID 30010440